CLINICAL TRIAL: NCT02874833
Title: The Efficacy of Exercise in Depressive Episodes of Unipolar Depression and Bipolar Affective Disorders
Brief Title: Exercise for Depression
Acronym: EXDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Department of Psychiatry and Psychotherapy, University Medical Center, Mainz (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Perikles Simon, Professor for Sports Medicine MD PHD, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXDEP_1
Record Dates: First submitted 2016-08-08; First posted 2016-08-22 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Depression, Unipolar; Bipolar Disorder
Keywords: Depression; Unipolar depression; Bipolar affective disorder; Exercise; Internet-based intervention
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Group (Experimental): Experimental arm type will assess whether a newly developed, supervised 8-week individualized, internet-based exercise therapy is effective in reducing depressive symptoms.
  Interventions: Other: Exercise
- Treatment as usual group (No Intervention): Treatment as usual. Other form of therapy (e.g. antidepressive medication) will not be affected.

INTERVENTIONS:
Other: Exercise — After performance diagnostics, participants will complete an 8-week supervised, individualized exercise program. Training will include up to 3 aerobic training sessions and up to two resistance training units per week.
  Arms: Exercise Group

SUMMARY:
A randomized single-blinded prospective study to evaluate the efficacy of an individualized supervised 8-week exercise program in subjects with moderate to severe depressive episodes compared to treatment-as-usual

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of a supervised and indvidualized 8-week exercise program compared to treatment-as-usual in subjects with a moderate or severe depressive episode in the context of unipolar depression or bipolar affective disorders. Numerous previous studies suggest that exercise may help to improve the symptoms of depression. Moreover, exercise was shown to enhance neuroplasticity in adults whereas depression results in decreased neuroplasticity. Here, we aim at elucidating whether a newly developed supervised, Internet-based, individualized exercise program of the Institute of Sports Science and the Department of Psychiatry and Psychotherapy at the University Mainz is more effective in reducing depressive symptoms than treatment-as-usual. Furthermore, this study will clarify if severely depressed subjects are able to adhere to an internet-based exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations.
2. Aged 18 to 65 years old, inclusive, at the time of informed consent.
3. Montral Cognitive Assessment (MoCA) > 26 to exclude cognitive impairment.
4. Apart from a clinical diagnosis of major depression or bipolar affective disorder, the subject must be in good health as determined by the Investigator, based on medical history and physical examination.
5. QIDS scores > 5

Exclusion Criteria:

1. Use of antidepressive medications or benzodiazepines at doses that have not been stable for at least 6 weeks prior to Screening
2. Psychotherapy that started less than 8 weeks prior to Screening
3. Any clinically significant psychiatric illness other than major depression or bipolar affective disorder
4. Transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to Screening
5. Any uncontrolled medical or neurological/neurodegenerative condition that, in the opinion of the Investigator, might impair treatment compliance and adherence
6. History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class III or IV), or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to Screening
7. Clinically significant 12-lead ECG abnormalities, as determined by the Investigator
8. Uncontrolled hypertension defined as: average of 3 systolic blood pressure [SBP]/diastolic blood pressure [DBP] readings > 165/100 mmHg at Screening
9. History of malignancy or carcinoma, with the following exceptions:

   i) Subjects with cancers in remission more than 5 years prior to Screening. ii) Subjects with a history of excised or treated basal cell or squamous carcinoma. iii) Subjects with prostate cancer in situ.
10. History of seizure within 2 years prior to Screening.
11. Recent history (within 1 year of Screening) of alcohol or substance abuse as determined by the Investigator, a positive urine drug (due to non-prescription drug) or alcohol test at Screening
12. Clinically significant systemic illness or serious infection (e.g., pneumonia, septicemia) within 30 days prior to or during Screening
13. History of human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV)
14. Any other medical conditions (e.g., renal disease) that are not stable or controlled, or, which in the opinion of the Investigator, could affect the subject's safety or interfere with the study assessments
15. Female subjects who are pregnant or currently breastfeeding
16. Participation in another study
17. Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the subject unsuitable for enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Severity of depressive symptoms - Quick Inventory of Depressive Symptomatology - clinical rating-16 (QIDS C-16) | 8 weeks
  Change of Score on the QIDS C-16 after 8 weeks compared to baseline.
Severity of depressive symptoms - Quick Inventory of Depressive Symptomatology - self-report-16 (QIDS SR-16) | 8 weeks
  Change of Score on the QIDS SR-16 after 8 weeks compared to baseline.

SECONDARY OUTCOMES:
Adherence of internet-based concept | 8 weeks
  Adherence of internet-based concept using an own questionnaire. Participants respond at the end of every week how they managed their individualized exercise schedule in terms of number of realised training sessions, average heart rate and subjective perceived exertion.
Placebo effect of exercise (QIDS-SR16) | 8-10 days
  Change of Score on the QIDS-SR16 after one week of training to determine placebo effect of exercise.
Placebo effect of exercise (QIDS-C16) | 8-10 days
  Change of Score on the QIDS-C16 after one week of training to determine placebo effect of exercise.
Peak oxygen uptake (VO2peak) | 8 weeks
  Change of VO2peak after 8 weeks compared to baseline. Participants will be subjected to a step-wise treadmill test at baseline and after 8 weeks.
Lactate threshold | 8 weeks
  Change of lactate threshold using the baseline +1.5 mmol model after 8 weeks compared to baseline.
Short form 36 (SF36) health survey questionnaire | 8 weeks
  Change of score on the SF-36 after 8 weeks compared to baseline.
General self efficacy questionnaire (GSE) | 8 weeks
  Change of score on the GSE after 8 weeks compared to baseline.
Global Clinical Issues (GCI) | 8 weeks
  Change of score on GCI after 8 weeks compared to baseline.
Circulating, cell-free DNA (cfDNA) | 8 weeks
  Change of cfDNA concentrations after 8 weeks compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Jung, PD Dr. habil., Principal Investigator — Department of Psychiatry and Psychotherapy, University Medical Center, Mainz
Locations (2):
- Germany (2):
  - Department of Psychiatry and Psychotherapy, University Medical Center, Mainz, Mainz, Rhineland-Palatinate
  - Department of Sports Medicine, Johannes Gutenberg University, Mainz, Mainz, Rhineland-Palatinate

REFERENCES:
- [Background] Cooney GM, Dwan K, Greig CA, Lawlor DA, Rimer J, Waugh FR, McMurdo M, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD004366. doi: 10.1002/14651858.CD004366.pub6. PMID 24026850
- [Background] Malykhin NV, Coupland NJ. Hippocampal neuroplasticity in major depressive disorder. Neuroscience. 2015 Nov 19;309:200-13. doi: 10.1016/j.neuroscience.2015.04.047. Epub 2015 Apr 28. PMID 25934030
- [Background] van Praag H, Shubert T, Zhao C, Gage FH. Exercise enhances learning and hippocampal neurogenesis in aged mice. J Neurosci. 2005 Sep 21;25(38):8680-5. doi: 10.1523/JNEUROSCI.1731-05.2005. PMID 16177036
- [Background] Yau GS, Lee JW, Woo TT, Wong RL, Wong IY. Central Macular Thickness in Children with Myopia, Emmetropia, and Hyperopia: An Optical Coherence Tomography Study. Biomed Res Int. 2015;2015:847694. doi: 10.1155/2015/847694. Epub 2015 Jun 8. PMID 26167504
- [Derived] Haller N, Lorenz S, Pfirrmann D, Koch C, Lieb K, Dettweiler U, Simon P, Jung P. Individualized Web-Based Exercise for the Treatment of Depression: Randomized Controlled Trial. JMIR Ment Health. 2018 Oct 12;5(4):e10698. doi: 10.2196/10698. PMID 30314962
- [Derived] Pfirrmann D, Haller N, Huber Y, Jung P, Lieb K, Gockel I, Poplawska K, Schattenberg JM, Simon P. Applicability of a Web-Based, Individualized Exercise Intervention in Patients With Liver Disease, Cystic Fibrosis, Esophageal Cancer, and Psychiatric Disorders: Process Evaluation of 4 Ongoing Clinical Trials. JMIR Res Protoc. 2018 May 22;7(5):e106. doi: 10.2196/resprot.8607. PMID 29789277